CLINICAL TRIAL: NCT02706444
Title: A Prospective, Multicenter, Randomized, Controlled Trial for Comparison of Drug-coated Balloon Versus Conventional Balloon Angioplasty in Venous Anastomotic Stenosis of Hemodialysis Graft
Brief Title: Drug-coated Balloon Versus Conventional Balloon Angioplasty in Hemodialysis Graft
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang Woo Park, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH1140101
Record Dates: First submitted 2015-11-05; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Vascular Graft Anastomotic Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Balloon Angioplasty (Active Comparator): Conventional balloon angioplasty. After fistulogram, full expansion of conventional balloon catheter under fluoroscopy guidance in > 50% venous anastomotic stenosis of hemodialysis graft and ≦4cm from venous anastomosis site in lesion length, confirmed by fistulogram
  Interventions: Device: Conventional Balloon angioplasty
- Drug-Coated Balloon Angioplasty (Active Comparator): Drug-coated balloon angioplasty. After fistulogram, full expansion of drug-coated balloon catheter under fluoroscopy guidance in > 50% venous anastomotic stenosis of hemodialysis graft and ≦4cm from venous anastomosis site in lesion length, confirmed by fistulogram
  Interventions: Device: Drug-coated Balloon angioplasty

INTERVENTIONS:
Device: Conventional Balloon angioplasty — After fistulogram, full expansion of drug-coated balloon catheter under fluoroscopy guidance in > 50% venous anastomotic stenosis of hemodialysis graft and ≦4cm from venous anastomosis site in lesion length, confirmed by fistulogram. Then, participants were divided into two groups (Conventional balloon angioplasty or Drug-coated balloon angioplasty)
  Arms: Conventional Balloon Angioplasty
Device: Drug-coated Balloon angioplasty — After fistulogram, full expansion of drug-coated balloon catheter under fluoroscopy guidance in > 50% venous anastomotic stenosis of hemodialysis graft and ≦4cm from venous anastomosis site in lesion length, confirmed by fistulogram. Then, participants were divided into two groups (Conventional balloon angioplasty or Drug-coated balloon angioplasty)
  Arms: Drug-Coated Balloon Angioplasty

SUMMARY:
To evaluate the role of DCB angioplasty for venous anastomotic stenosis of hemodialysis graft, investigators would like to perform randomized study comparing the results of drug- coated balloon angioplasty with conventional balloon angioplasty in the treatment in venous anastomotic stenosis of AVG in terms of patency.

DETAILED DESCRIPTION:
Study Procedure The Interventional angiographic suit will follow the standard hemodialysis related interventional procedure for PTA. Fistulogram will be performed prior to PTA. All enrolled patients should undergo 3 and 6-month follow-up fistulogram and information will be collected and recorded on the treated study vessel and pictures through angiographic image. These data will be recorded on clinical recording form using an excel program.

1. Pretreatment evaluation 1.1 All procedures will be performed after obtaining written informed consent from patients. No specific pre-treatment regimen will be needed.

   1.2 After sterile preparation and draping, percutaneous access will be gained in an appropriately chosen hemodialysis graft after application of local anesthesia. Diagnostic fistulogram was performed to identify and evaluate the target lesion and any possible secondary lesions. In case of thrombotic occlusion of AVG, diagnostic fistulogram will be done after successful aspiration thrombectomy though a sheath.

   1.3 All lesions were characterized by location, length, and degree of stenosis. The degree of stenoses was evaluated in two orthogonal planes, and the greatest degree of stenoses was used for subsequent anatomic measurements. Anatomic measurements were made with use of a calibrated reference marker or software within the angiographic imaging system. The reference vessel was defined as an adjacent segment of normal vein or graft located adjacent to the target lesion. The degree of stenosis was reported as the maximum diameter reduction compared with the reference vessel diameter.
2. PTA in venous anastomosis of AVG 2.1 Vascular sheaths will be used in all cases. 2.2 Balloon diameter will be chosen at the operator's discretion, generally starting with a balloon 10% oversized compared with the adjacent normal vein or graft in both groups (Reference Vessel Diameter: RVD).

   2.3 Balloon length will be also chosen at the discretion of the operator: In general, 4-cm- or 6cm-long balloons can be used for some long lesions.

   2.4 If patient requested the sedation, conscious sedation can be done. 2.5 After crossing the stenosis with a guide wire, the conventional balloon catheter was appropriately positioned across the lesion under fluoroscopic guidance. With the use of an inflation device with a pressure gauge, the balloon catheter was gradually inflated until the stenosis was eliminated.

   2.6 Randomization will be assigned after successful conventional balloon angioplasty in venous anastomotic stenosis of AVG. After conventional angioplasty, patients will be randomly assigned to undergo DEB angioplasty or to receive conventional balloon angioplasty for 3 minutes (upto norminal pressure).

   2.7 If the patient will be randomly assigned to the DEB group, an In.Pact® Drug-eluting balloon catheter (6, 7mm in diameter, ≦6cm in length) will be used in addition to conventional balloon angioplasty. A balloon diameter and length will be equal to that used in the conventional balloon angioplasty group.
3. Procedure Materials PRODUCT SIZE LENGTHS Drug Eluting balloon In.Pact® 6,7mm 4, 6cm Conventional balloon Various conventional balloon catheter 6,7mm 4, 6cm
4. Follow-up

   * All patients will be followed after PTA. When patients visit hemodialysis unit 3 and 6 months after PTA, the patient's record will be updated.
   * All patients that visit hemodialysis unit will be brought to angiographic suit to undergo follow-up fistulogram and evaluate the re-stenosis.
   * Clinical follow-up will be performed in hemodialysis unit, including checking the status of hemodialysis using a those circuits and general work-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age of more than 19
2. Hemodialysis patients with AVG in their arms: Graft should be implanted 30 days ago before enrollment
3. Vascular access actively used for hemodialysis: At least one hemodialysis successful session before enrollment.
4. Clinical signs of access dysfunction: decreased thrill, increased pulsatility, development collateral veins, limb swelling, difficulty in cannulation, prolonged bleeding after hemodialysis, high venous pressure or decreased hemodialysis flow rate during hemodialysis.
5. > 50% venous anastomotic stenosis of AVG, confirmed by fistulogram (angiography).
6. ≦ 4cm from venous anastomosis site in lesion length
7. Reference diameter < 7mm of non-stenotic vessel or graft adjacent to venous stenosis.
8. Full expansion of conventional balloon during primary balloon angioplasty, confirmed by fluoroscopy.

Exclusion criteria

1. Patients unable to provide informed consent
2. Patient unable to abide with study follow-up protocol.
3. Patient participating in other relevant or conflicting studies
4. Bare metal stent or stent-graft placed previously
5. Hemodynamically significant stenosis of the central venous system
6. ≧50% stenosis in arterial anastomotic site or venous outflow tract, non including venous anastomosis site
7. Stenosis with a corresponding thrombosis treated within 7 days before enrollment.
8. Limited life expectancy less than 6 months
9. Sepsis or active infection.
10. Recent arm thrombophlebitis (< 6months).
11. Allergy or other known contraindication to iodinated contrast media, heparin, or paclitaxel
12. Pregnancy or Nursing state

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Primary patency (Fistulogram can be used for measurement of stenosis) | 6 months

IPD SHARING:
Plan to Share IPD: No